CLINICAL TRIAL: NCT06811623
Title: Omentopexy After Sleeve Gastrectomy in Children and Adolescences, is it Effective in Reducing Post-operative Complications.
Brief Title: Omentopexy After Sleeve Gastrectomy in Children and Adolescences.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Daboos (Other)
Responsible Party: Sponsor-Investigator, Mohammad Daboos, Professor at Pediatric Surgery Department, Al-Azhar University., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2015OBSGN63
Record Dates: First submitted 2025-01-26; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Morbid Obesity; Pediatric Obesity; LAP
MeSH Terms: conditions — Obesity, Morbid; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: group 1: included 24 patients managed with Laparoscopic Sleeve Gastrectomy with omentopexy and group 2: included 24 patients managed with Laparoscopic Sleeve Gastrectomy without omentopexy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with Omentopexy (Active Comparator): Laparoscopic Sleeve Gastrectomy with omentopexy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy with omentopexy
- Group without Omentopexy (Active Comparator): Laparoscopic Sleeve Gastrectomy without omentopexy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy without omentopexy

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy with omentopexy — Laparoscopic Sleeve Gastrectomy with omental fixation to the gastric tube
  Arms: Group with Omentopexy
Procedure: Laparoscopic Sleeve Gastrectomy without omentopexy — Laparoscopic Sleeve Gastrectomy without omental fixation to the gastric tube
  Arms: Group without Omentopexy

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is a restrictive bariatric operation, has become one of the most commonly performed bariatric surgeries. Postoperative gastrointestinal complications are agonizing in patients underwent this procedure. Most of these complications can be prevented by omentopexy in association with sleeve gastrectomy. The Primary aim of this study to assess the effectiveness of omentopexy during laparoscopic sleeve gastrectomy in reducing post-operative complication.

DETAILED DESCRIPTION:
This study was a carried out as a prospective study of 48 patients with obesity between January 2015 and October 2024. The patients were divided into 2 groups; group 1: included 24 patients managed with LSG with omentopexy and group 2: included 24 patients managed with LSG without omentopexy. Pre- operation data and post operation outcomes were taken for all patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of 40 kg/m2 or
* BMI of 35 kg/m2 due to at least 1 comorbid condition

Exclusion Criteria:

* secondary obesity
* more than 18 years
* previous operation

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
post-operative complications | 6 months
  post operative nausea, vomiting and leakage

SECONDARY OUTCOMES:
operative time and hospital stay | 6 months
  the length of operative procedure and post-operative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Daboos, Principal Investigator — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No